CLINICAL TRIAL: NCT02111447
Title: Post Anesthesia Emergence and Behavioral Changes in Children Undergoing MRI: Comparative Study Using Propofol, Sevoflurane and Isoflurane
Brief Title: Post Anesthesia Emergence and Behavioral Changes in Children Undergoing MRI
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Not enough participants
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Jerrold Lerman, Clinical Professor of Anesthesiology, State University of New York at Buffalo
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 412889-6
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Delirium on Emergence
Keywords: children; sevoflurane; isoflurane; propofol; anesthesia; MRI; delirium
MeSH Terms: conditions — Emergence Delirium; Delirium | interventions — Propofol; Sevoflurane; Isoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sevoflurane, propofol, Nasal oxygen (Active Comparator): After securing the IV, sevoflurane will be discontinued and a propofol infusion will be started at the dose of 300 mcg/kg/min depending on the child's age and neurologic status. A bolus of propofol will not be administered. Oxygen will be delivered via nasal prongs at 2 liters per minute. The infusion rate of propofol will be decreased to 250 after 15 min and then 200 mcg/kg/min also after 15 min. Supplemental IV boluses of Propofol (0.5 mg/kg) will be administered if the child moves or if signs of light anesthesia are noticed. The propofol infusion may also be increased in response to light anesthesia.
  Interventions: Drug: Propofol
- Sevoflurane, Propofol, LMA (Active Comparator): After securing the IV, weight appropriate LMA will be inserted and sevoflurane will be discontinued and a propofol infusion will be started at the dose of 300 mcg/kg/min depending on the child's age and neurologic status. Oxygen in air will be delivered via LMA. The infusion rate of propofol will be decreased to 250 after 15 min and then 200 mcg/kg/min after another 15 min. Supplemental IV boluses of Propofol (0.5 mg/kg) will be given if the child moves or exhibits signs of light anesthesia. The propofol infusion may also be increased in response to light anesthesia.
  Interventions: Drug: Propofol; Drug: Sevoflurane
- Sevoflurane, sevoflurane, LMA (Active Comparator): After securing the IV, weight appropriate LMA will be inserted and sevoflurane continued at 3% inspired concentration. Oxygen in air will be delivered via LMA at 2 lpm. The sevoflurane may be increased or decreased in 0.5% increments as needed.
  Interventions: Drug: Sevoflurane
- Sevoflurane, isoflurane, LMA (Active Comparator): After securing the IV, weight appropriate LMA will be inserted , sevoflurane will be discontinued and isoflurane will be administered at 2 % inspired concentration. Oxygen in air will be delivered via LMA at 2 lpm. Isoflurane may be increased or decreased in 0.5% increments as needed.
  Interventions: Drug: Sevoflurane; Drug: Isoflurane

INTERVENTIONS:
Drug: Propofol — Propofol infusion with nasal oxygen
  Other Names: Diprivan 1%
  Arms: Sevoflurane, Propofol, LMA; Sevoflurane, propofol, Nasal oxygen
Drug: Propofol — Propofol infusion with an LMA
  Other Names: 1% Diprivan
  Arms: Sevoflurane, propofol, Nasal oxygen
Drug: Sevoflurane — Sevoflurane with an LMA
  Other Names: Sevorane
  Arms: Sevoflurane, Propofol, LMA; Sevoflurane, isoflurane, LMA; Sevoflurane, sevoflurane, LMA
Drug: Isoflurane — Isoflurane with an LMA
  Other Names: Forane
  Arms: Sevoflurane, isoflurane, LMA

SUMMARY:
Children who receive general anesthesia may become agitated (emergence delirium) in the recovery period. This occurs more often after inhalational anesthetics, particularly sevoflurane and desflurane than after propofol. However, agitation after anesthesia in children may be difficult to distinguish from pain; accordingly studies are ideally designed during MRI to obviate the contribution of pain during emergence. Airway complications have been reported after LMA and isoflurane more commonly than with IV propofol and nasal prongs. Whether the airway complications were due to the LMA or the isoflurane was unclear. Therefore, this study was designed to study the incidence of 1. agitation after sevoflurane compared with IV propofol and 2. airway complications after LMA or nasal prongs.

DETAILED DESCRIPTION:
180 children, ASA physical status 1 or 2 will be recruited for elective MRI scan. Randomized after consent is obtained to one of four groups. Anxiety will be assessed preoperatively using the modified Yale preoperative anxiety scale. Children will be accompanied by one parent to MRI scanner where monitors are applied. All children will have anesthesia induced with nitrous oxide and oxygen followed by sevoflurane until IV is established. Thereupon, they will be managed by their randomization assignment. The propofol pump will be concealed at all times. If propofol was used, it will be disconnected from the patient and residual propofol in the line flushed so prevent unblinding the patient's assignment. A blinded observer will be present to evaluate the patient when emergence begins. The single blinded observer will follow the patient from the MRI scanner through recovery room evaluating vital signs as well as emergence delirium (using the PAED scale). A PAED score > 12 at any time during emergence period will confirm the diagnosis of emergence delirium. After discharge from hospital, a post-discharge questionnaire will be completed at 12, 24 and 48 hours after discharge. All parents will be called to retrieve the questionnaire results after 48 hours after discharge from hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-12yrs,
* ASA Class I-II,
* Fasting,
* Unmedicated,
* Elective MRI scan

Exclusion Criteria:

* Cognitive impairment,
* On psychotropic medications,
* Taking multiple (>2) antiepileptic medications,
* Requiring endotracheal intubation for GA

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerrold Lerman, MD, Principal Investigator — Women And Childrens Hospital Of Buffalo; Christopher Heard, MD, Principal Investigator — Women And Childrens Hospital Of Buffalo
Locations (1):
- Women and Chidren's Hospital Of Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sevoflurane, Propofol, Nasal Oxygen | Sevoflurane, Propofol, LMA | Sevoflurane, Sevoflurane, LMA | Sevoflurane, Isoflurane, LMA
Started | 0 | 5 | 1 | 0
Completed | 0 | 5 | 1 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: start study
Groups:
- Total: Total of all reporting groups
Arm/Group | Sevoflurane, Propofol, Nasal Oxygen | Sevoflurane, Propofol, LMA | Sevoflurane, Sevoflurane, LMA | Sevoflurane, Isoflurane, LMA | Total
Number analyzed (Participants) | 0 | 5 | 1 | 0 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 5 | 1 | 0 | 6
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 3 | 0 |  | 3
  Male |  | 2 | 1 |  | 3
Region of Enrollment [Number; unit: participants]
  United States |  | 5 | 1 |  | 6

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Delirium on Emergence
Description: Delirium on emergence will be assessed using the PAED scale by a blinded observer in the post anesthesia period. A score >12 constitutes a diagnosis of delirium in children. The post anesthesia period is usually <2 hours after anesthesia.
Time Frame: WIthin 2 hours of emergence from anesthesia
Population: none recruited that that group
Measure: Count of Participants; unit: Participants
Arm/Group | Sevoflurane, Propofol, Nasal Oxygen | Sevoflurane, Sevoflurane, LMA | Sevoflurane, Propofol, LMA | Sevoflurane, Isoflurane, LMA
Number analyzed (Participants) | 0 | 1 | 5 | 0
Participants | 0 | 1 | 5 | 0

2. Secondary Outcome: Incidence of Airway Complications
Description: All airway reflex responses including airway obstruction breath holding, coughing, laryngospasm, desaturation <92% for >15 s regardless of the cause, bronchospasm, secretions and hiccups
Time Frame: WIthin 2 hours of emergence from anesthesia
Population: none recruited to that group
Measure: Count of Participants; unit: Participants
Arm/Group | Sevoflurane, Propofol, Nasal Oxygen | Sevoflurane, Sevoflurane, LMA | Sevoflurane, Propofol, LMA | Sevoflurane, Isoflurane, LMA
Number analyzed (Participants) | 0 | 1 | 5 | 0
Participants | 0 | 1 | 5 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: Definition does not differ.
Arm/Group | Sevoflurane, Propofol, Nasal Oxygen | Sevoflurane, Sevoflurane, LMA | Sevoflurane, Propofol, LMA | Sevoflurane, Isoflurane, LMA
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1 | 0/5 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/5 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/5 | 0/0

LIMITATIONS AND CAVEATS:
none study not completed due to facility issues

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No